CLINICAL TRIAL: NCT06124300
Title: A Single Group Study to Evaluate the Effects of a Female Hormone Balance Supplement on Symptoms of Polycystic Ovary Syndrome and Severe Premenstrual Syndrome
Brief Title: Effects of a Female Hormone Balance Supplement on Symptoms of Polycystic Ovary Syndrome and Severe Premenstrual Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rael (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20336
Record Dates: First submitted 2023-11-04; First posted 2023-11-09 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Polycystic Ovary Syndrome; Premenstrual Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome; Premenstrual Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Female Hormone Balance Supplement (Experimental): Participants will add 1 scoop of the powder to a drink of choice every morning.
  Interventions: Dietary Supplement: Female Hormone Balance Supplement

INTERVENTIONS:
Dietary Supplement: Female Hormone Balance Supplement — The product contains: Myo-Inositol D-Chiro Inositol Folic Acid Vitamin D Vitamin B12

SUMMARY:
This is a virtual single group study that will last 12 weeks. Participants will take 1 scoop of the female hormone balance supplement, and mix it with their drink of choice every morning. Questionnaires will be completed at baseline, 1 week, 2 weeks, 4 weeks, and 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 - 55
* BMI less than 35
* Self-reported concerns around irregular menstrual cycles and ovulation, mood swings, stress, irritability, and low energy
* Generally healthy - don't live with any uncontrolled chronic disease
* Self-reported symptoms of PCOS - irregular periods
* Self-reported concerns with hormonal skin issues

Exclusion Criteria:

* Anyone with pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders
* Anyone with known severe allergic reactions
* Anyone who is pregnant, breastfeeding, or attempting to become pregnant
* Unwilling to follow the study protocol

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Changes in menstrual cycle regularity. | Baseline to Week 12
  Study-specific questionnaires completed by participants. Questionnaires utilize a 5-point Likert scale with 5 representing the most favorable/best outcome (e.g., "Very regular") and 1 representing the least favorable/worst outcome (e.g., "Extremely irregular").
Changes in hormonal acne. | Baseline to Week 12
  Study-specific questionnaires completed by participants. Questionnaires utilize a 5-point Likert scale with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").
Changes in skin issues throughout the menstrual cycle. | Baseline to Week 12
  Study-specific questionnaires completed by participants. Questionnaires utilize a 5-point Likert scale with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").

SECONDARY OUTCOMES:
Changes in overall mood. | Baseline to Week 12
  Study-specific questionnaires completed by participants. Questionnaires utilize a 5-point Likert scale with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").
Changes in stress levels. | Baseline to Week 12
  Study-specific questionnaires completed by participants. Questionnaires utilize a 5-point Likert scale with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").
Changes in food cravings. | Baseline to Week 12
  Study-specific questionnaires completed by participants. Questionnaires utilize a 5-point Likert scale with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").
Changes in energy. | Baseline to Week 12
  Study-specific questionnaires completed by participants. Questionnaires utilize a 5-point Likert scale with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").
Changes in menstrual cramps. | Baseline to Week 12
  Study-specific questionnaires completed by participants. Questionnaires utilize a 5-point Likert scale with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided